CLINICAL TRIAL: NCT02536027
Title: Effect of Continuous Venovenous Hemofiltration on the Plasma Level of Neutrophil Gelatinase-associated Lipocalin in Critical Ill Patients With Septic Acute Kidney Injury
Brief Title: Effect of CVVH on NGAL in Septic AKI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First People's Hospital of Chenzhou (Other)
Responsible Party: Principal Investigator, Xingui Dai, Critical Care Medicine, First People's Hospital of Chenzhou
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: FirstHospitalchenzhou
Record Dates: First submitted 2015-08-20; First posted 2015-08-31 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Acute Kidney Injury
Keywords: continuous venovenous hemofiltration; neutrophil gelatinase-associated lipocalin; sepsis; acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury; Sepsis | interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- septic AKI patients (Experimental): septic AKI patients requiring CVVH
  Interventions: Procedure: continuous venovenous hemofiltration

INTERVENTIONS:
Procedure: continuous venovenous hemofiltration — Continuous renal replacement therapy (CRRT) has become routine for patients with AKI, chronic renal failure, ﬂuid overload as well as oliguria in ICU. In clinical practice, continuous venovenous hemofiltration (CVVH) is actually the method of choice for CRRT in critically ill and hemodynamic instable patients. CVVH has significant beneficial effects on removing inflammatory cytokines, improving oxygen index, decreasing vasopressor requirements, increasing cardiac index, and regulating immune dysfunction, specifically in patients with septic shock.
  Other Names: continuous renal replacement therapy

SUMMARY:
The plasma level of neutrophil gelatinase-associated lipocalin (NGAL) in critically ill patients with AKI is not affected by continuous venovenous hemofiltration (CVVH). However, it remains unclear if this also applies to sepsis-induced AKI, as considerable evidence suggests that the pathophysiology of septic AKI is different from other causes of AKI.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is an increasingly common and potentially catastrophic complication in critically ill patients. The incidence of AKI increases in recent years; about half of all patients in the intensive care units (ICU) develop AKI. AKI is associated with a significantly increased length of hospital stay and high mortality rates. Approximately, 50% of AKI is induced by sepsis.

Continuous renal replacement therapy (CRRT) has become routine for patients with AKI, chronic renal failure, ﬂuid overload as well as oliguria in ICU. In clinical practice, continuous venovenous hemofiltration (CVVH) is actually the method of choice for CRRT in critically ill and hemodynamic instable patients. CVVH has significant beneficial effects on removing inflammatory cytokines, improving oxygen index, decreasing vasopressor requirements, increasing cardiac index, and regulating immune dysfunction, specifically in patients with septic shock. So far, there is no uniform standard to define the timing of discontinuation of CRRT for AKI, as predicting recovery of renal function in patients with AKI during CRRT is difficult. The Beginning and Ending Supportive Therapy for the Kidney (BEST Kidney) study suggested the urinary output > 500ml per day as the predictor for successful discontinuation of CRRT. However, the urinary output is often affected by clinical interventions (e.g. using diuretics). Thus, it is of great importance to find out a reliable biomarker to reflect the renal function of the patients who receiving CRRT. Cystatin (Cys) C has received the most interest in previous studies. The results showed serum Cys C concentrations were declined in different types of RRT (including intermittent hemodialysis and CVVH). This indicates Cys C is unfit as an indicator for persistent renal injury or renal recovery in critically ill patients during CRRT.

Neutrophil gelatinase-associated lipocalin (NGAL), a 25-kDa protein that covalently binds to gelatinase from neutrophils, is generally expressed at very low levels in several human tissues, however, in case of ischemia, infection, or toxic damage, NGAL rapidly released by activated neutrophils. Numerous studies have confirmed NGAL as a better indicator of AKI than serum creatinine (SCr). Schilder and colleagues reported that the plasma level of NGAL in critically ill patients with AKI is not affected by continuous venovenous hemofiltration (CVVH). However, it remains unclear if this also applies to sepsis-induced AKI, as considerable evidence suggests that the pathophysiology of septic AKI is different from other causes of AKI.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive adult (>18 years) patients with septic AKI undergoing CRRT

Exclusion Criteria:

* those with end-stage renal disease
* those who had undergone renal transplant
* those with cancer
* those who had contracted acquired immunodeficiency syndrome
* those who had undergone high-dose steroid treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
plasma level of neutrophil gelatinase-associated lipocalin | 0-12 hours
  The specimens in the inlet, outlet and ultrafiltrate were obtained at the beginning of CVVH (T0) and 2 h (T2h), 4 h (T4h), 8 h (T8h), and 12 h (T12h) after setup of continuous renal replacement therapy (CRRT).The plasmatic NGAL level was measured with enzyme-linked immunosorbent assay (R&D Systems, UK, Lipocalin2/NGAL Duoset, DY1757).

CONTACTS AND LOCATIONS:
Overall Officials: Dixian DX Luo, MS, Study Director — Chenzhou First people Hospital

REFERENCES:
- [Derived] Dai X, Li T, Zeng Z, Fu C, Wang S, Cai Y, Chen Z. The effect of continuous venovenous hemofiltration on neutrophil gelatinase-associated lipocalin plasma levels in patients with septic acute kidney injury. BMC Nephrol. 2016 Oct 19;17(1):154. doi: 10.1186/s12882-016-0363-y. PMID 27760529